CLINICAL TRIAL: NCT05230433
Title: Implications of Insulin Resistance and Cardiorespiratory Fitness in the Metabolic Response to a High-fat Meal Challenge in Pediatrics
Brief Title: High-fat Meal Challenge in Pediatrics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jennifer L. Meijer, Principal Investigator; Scientist, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY02001316
Record Dates: First submitted 2022-01-06; First posted 2022-02-09 (Actual); Results first posted 2025-07-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Pediatric Obesity; Insulin Resistance
MeSH Terms: conditions — Pediatric Obesity; Insulin Resistance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High-fat Metabolic Challenge (Experimental): Participants will consume a high-fat agent one time, at the second study visit.
  Interventions: Dietary Supplement: High-fat Challenge

INTERVENTIONS:
Dietary Supplement: High-fat Challenge — The shake will be composed of a mixture of BOOST Glucose Control(R) (Nestlé Products) supplemented with palm oil. Each participant will consume a volume of liquid equivalent to 25% of their estimated daily caloric needs, calculated by the USDA Dietary Reference Intakes using a moderate activity factor.

SUMMARY:
The objective is to determine if how physical fitness, measured using a treadmill maximal oxidative capacity test, is associated with the capacity to metabolize a high-fat meal in pediatrics (ages 8-17 years). Ability to metabolize the meal will be assessed by profiling mitochondrial and extra-mitochondrial fatty acid metabolites. The investigators will test if fatty acid oxidation mediates the relationship between fitness and markers of metabolic health, such as insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 8-17 years with a BMI-percentile ≥ 5th.

Exclusion Criteria:

* Previous diagnosis of type 1 or 2 diabetes.
* Use of concurrent medications known to affect glucose metabolism (metformin, oral steroids, sulfonylureas, insulin).
* Evidence of inherited disorders of lipid metabolism.
* Inability to participant in the maximal aerobic capacity test on the treadmill.
* Allergies to palm oils or protein types within high-fat challenge, such as lactose and soy.
* Individuals who cannot speak and/or write in English.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Health, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was completed in September 2022 (n=15). Recruitment followed D-H IRB approval. Adolescents (8-17 years) were recruited through the Children's Hospital at Dartmouth Hitchcock (assisted by Dr. Susanne Tanski), the Weight and Wellness Center (assisted by Dr. Auden McClure), and, as needed, through the community. Flyers have been developed by DHMC marketing.
Pre-assignment Details: No pre-assignment occurred.
Groups:
- High-fat Metabolic Challenge: All participants consumed a high-fat agent at the second study visit. The shake was be composed of a mixture of BOOST Glucose Control(R) (Nestlé Products) supplemented with palm oil. Each participant will consume a volume of liquid equivalent to 25% of their estimated daily caloric needs, calculated by the USDA Dietary Reference Intakes using a moderate activity factor.
Period: Overall Study
Arm/Group | High-fat Metabolic Challenge
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | High-fat Metabolic Challenge
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 14 (3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 22.7 (6.1)

OUTCOME MEASURES:

1. Primary Outcome: Palatability of the High Fat Agent.
Description: Determine the number of participants that complete at least 75% of the shake (by weight).
Time Frame: 10 minutes
Measure: Count of Participants; unit: Participants
Groups:
- High-fat Metabolic Challenge: All participants consumed the high-fat challenge
Arm/Group | High-fat Metabolic Challenge
Number analyzed (Participants) | 15
Participants | 13
Statistical Analysis 1: Comparison: High-fat Metabolic Challenge; High fat agents were weighed pre- and post- providing the shake to the participant. All containers were tared to take into account straw, lid, and glass weight. Percentage of high-fat challenge consumed was calculated by post-shake weight / pre-shake weight. 13 out of 15 partcipants drank >75% of the shake; Test type: Other; p = 0.15, Chi-squared — p-value was not adjusted for multiple comparisons; Percent Consumed = 86

2. Secondary Outcome: BMI Percentile
Description: BMI percentile calculated for each participant. Average and standard deviations were reported.
Time Frame: At baseline
Measure: Mean (Standard Deviation); unit: percentile
Arm/Group | High-fat Metabolic Challenge
Number analyzed (Participants) | 15
percentile | 70 (24)
Statistical Analysis 1: Comparison: High-fat Metabolic Challenge; Fold change from 60 to 180 minutes of average medium chain acylcarnitine was calculated for each participant. Pearson correlation between BMI percentile and fold change was calculated; Test type: Other — No test vs. control groups; p = 0.65, Pearson Correlation — This p-value is not adjusted for multiple comparisons; Pearson Correlation between both secondary outcomes reported: BMI percentile and fold change between acylcarnitine at 60 minutes and 180 minutes post the high fat challenge

3. Secondary Outcome: Medium Chain Acylcarnitine Concentration
Description: Medium chain acylcarnitines profiled in the plasma include acylcarnitine 6:0, 8:0, 10:0, 10:1, 12:0, and 12:1. Medium chain acylcarntine concentration was averaged in each participant. Average and standard deviations were reported.
Time Frame: 60 and 180 minutes post consumption of high fat shake
Measure: Mean (Standard Deviation); unit: mircoM
Arm/Group | High-fat Metabolic Challenge
Number analyzed (Participants) | 15
mircoM
  Average MC acylcarnitine at 60 minutes | 0.055 (0.015)
  Average MC acylcarnitine at 180 minutes | 0.061 (0.014)

4. Secondary Outcome: Fold Change of Medium Chain Acylcarnitine at 60 and 180 Minutes.
Description: as for outcome 3
Time Frame: 60 and 180 minutes post consumption of high fat shake
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | High-fat Metabolic Challenge
Number analyzed (Participants) | 15
ratio | 0.902 (0.021)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from signing the consent document to 2 weeks post the high-fat challenge study visit. Participants concluded the study at this timepoint.
Description: No difference
Arm/Group | High-fat Metabolic Challenge
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/33/NCT05230433/Prot_SAP_000.pdf